CLINICAL TRIAL: NCT07132294
Title: Effects of Small-Sided Games Versus Sprint Interval Running on Aerobic Capacity and Training Load in Elite Football: A Randomized Controlled Trial
Brief Title: This Randomized Controlled Trial Investigated the Effects of Two Preseason Training Protocols-Small-sided Games (SSG) and Supramaximal Interval Running (SIR)-on Aerobic Capacity and Training Load in Elite Turkish Football Players. Forty Participants Were Randomly Assigned to Either Group, and Traini
Acronym: SIRvsSSG2023
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Hamza Kucuk, Associate professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKucuk-FootballTrial23; 76fb8a54f90e4d6c (Other: Cankiri Karatekin University Health Sciences Ethics Committee)
Record Dates: First submitted 2025-08-04; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Exercise Performance; Aerobic Capacity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supramaximal Interval Running (SIR (Experimental): Participants in this group performed supramaximal running intervals at 100-110% of their Maximal Aerobic Speed (MAS), three times per week for six weeks. The protocol consisted of 8 sets of maximal effort runs with passive recovery between bouts. Training progressed from 2-minute to 3-minute intervals during the study.
  Interventions: Behavioral: Exercise Intervention
- Supramaximal Interval Running (Experimental): A high-intensity interval running protocol designed to improve aerobic and anaerobic capacity in professional football players. Training intensities were based on each participant's MAS and progressed in duration and intensity throughout the 6-week preseason phase.
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — Supramaximal Interval Running (SIR) This protocol was individualized based on each player's Maximal Aerobic Speed (MAS). Training intensities were prescribed at 100% to 110% of each player's MAS. Each session consisted of eight sets. During the first three weeks, each set involved a 2-minute maximal effort run followed by 2 minutes of passive recovery. In the final three weeks, the duration of each set was extended to a 3-minute maximal run with 3 minutes of passive rest, increasing intensity and volume. SIR sessions were designed to enhance anaerobic capacity and lactate tolerance.
  Small-Sided Games (SSG) SSG sessions were implemented to develop agility, acceleration, tactical decision-making, and match-relevant conditioning. Training took place on regulation-size grass pitches, adjusted to maintain a consistent length-to-width ratio across all formats. Over the six-week intervention, game formats progressed from 4v4 to 7v7, with gradual increases in duration and pitch dimensions.
  Other Names: Structured Exercise Training

SUMMARY:
Purpose of the Study:

This study aimed to compare the physiological and performance-related effects of two different training methods in elite football players: supramaximal interval running (SIR) and small-sided games (SSG).

Who Can Participate:

Forty professional male football players (excluding goalkeepers) from the top two leagues in Turkey participated in this study. Participants were required to have no injuries or health problems that could affect their performance.

How the Study Will Work:

The study was conducted over a six-week preseason preparation period for the 2023-2024 season. Participants were randomly assigned to either the supramaximal interval running (SIR) group or the small-sided games (SSG) group. Both groups trained three times a week. Before and after the intervention, measurements such as maximal aerobic speed (MAS), total running distance, blood lactate levels, body composition (fat mass), and heart rate were taken.

Potential Benefits and Risks:

Both training approaches resulted in significant improvements in body weight, fat mass, running distance, and aerobic capacity. The information gained from this study could help determine the most effective training methods for elite football players. Since the study is similar to a standard training program, no serious risks are expected.

Results:

This study found that both supramaximal interval running (SIR) and small-sided games (SSG) training methods improved the physiological and performance outcomes of elite football players. However, the SIR protocol was found to be associated with more pronounced gains in aerobic capacity, anaerobic markers, and body composition. These findings emphasize the benefit of SIR during a short preseason preparation period. The results of the study can help in developing training programs tailored to individual needs and performance goals.

DETAILED DESCRIPTION:
Purpose of the Study:

The purpose of this study was to compare the physiological and performance-related effects of two different training methods in elite football players: supramaximal interval running (SIR) and small-sided games (SSG). The study specifically examined the concurrent effects of SIR and SSG within a structured off-season program.

Study Design:

This study employed a controlled, experimental pre-post-test design to compare the effects of SIR and SSG on physiological and performance outcomes in professional football players. Forty professional male outfield players from Türkiye's top two football leagues were randomly assigned to either the SIR or SSG groups. A six-week intervention was implemented during the preseason, with assessments conducted at baseline and post-intervention under standardized conditions.

Participants:

The study included 40 professional male football players from the Super League and the Trendyol 1st League in Turkey. Goalkeepers were excluded to ensure positional uniformity. Inclusion criteria were participation in at least 85% of scheduled training sessions, absence of musculoskeletal injuries or medical conditions affecting performance, and no use of medication or supplements influencing physiological responses.

Interventions:

SIR and SSG training were conducted three times per week over a six-week preseason period.

Supramaximal Interval Running (SIR):

SIR sessions were individualized based on each athlete's Maximal Aerobic Speed (MAS). The intensity was prescribed at 100% to 110% of each player's MAS, with each session consisting of eight sets. In the first three weeks, each set involved a 2-minute maximal effort run followed by 2 minutes of passive recovery. In the final three weeks, both intensity and duration were progressively increased, with each set extended to 3 minutes of maximal effort and 3 minutes of rest.

Small-Sided Games (SSG):

SSG sessions were implemented to develop agility, acceleration, tactical decision-making, and match-relevant conditioning. Over the six-week intervention, game formats progressed from 4v4 to 7v7, with gradual increases in duration and pitch dimensions to ensure a consistent training load. Each session consisted of four sets per game format, separated by 5-minute passive rest periods.

Measurements:

Assessments before and after the intervention included:

Body Composition: Body mass and fat mass were assessed using the InBody270 bioelectrical impedance analyzer.

Maximal Aerobic Speed (MAS): MAS was evaluated using a standardized 1,200-meter time trial.

Physiological and Performance Monitoring: Heart rate (HR) was continuously monitored using Polar H10 sensors. Internal training load was assessed using the Borg CR-10 scale for perceived exertion (RPE). Capillary blood samples were obtained post-session to measure blood lactate (LA) concentrations. Performance metrics were recorded with 50 Hz GPS devices and synchronized heart rate monitors.

ELIGIBILITY:
Inclusion Criteria:

* Professional male football players who are actively playing in the Super League and the 1st League of Turkey.

Between the ages of 18 and 30. Agree to participate in at least 85% of the scheduled training sessions.

Exclusion Criteria:

* Goalkeepers (to ensure positional uniformity). Presence of musculoskeletal injuries or medical conditions that could affect performance.

Use of any medication or supplements that could influence physiological responses.

Suffering an injury or illness during the study and failing to attend at least 85% of the training sessions.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Maximal Aerobic Speed (MAS) | Baseline and after 6 weeks
  Description: Measured using a 1,200-meter time trial on a natural grass pitch. Unit of Measure: meters/second (m/s)
Total Running Distance | Throughout the 6-week intervention
  Measured using 50 Hz GPS devices.

SECONDARY OUTCOMES:
Blood Lactate Concentration (LA) | Immediately post-training sessions during the intervention
  Description: Measured from fingertip capillary blood samples using Lactate Pro 2 analyzer.
  Unit of Measure: millimoles per liter (mmol/L)
Fat Mass | Time Frame: Baseline and after 6 weeks
  Measured using the InBody270 bioelectrical impedance analyzer. Unit of Measure: kilograms (kg)
Heart Rate (HR) | During training sessions across the 6-week period
  Measured continuously using Polar H10 heart rate sensors. Unit of Measure: beats per minute (bpm)
Rating of Perceived Exertion (RPE) | Immediately post-training sessions during the intervention
  Measured using the Borg CR-10 scale.
  Unit of Measure: CR-10 score (0-10 scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University, Atakent, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Upon publication of the primary manuscript, the individual participant data (IPD) will be made available upon request to qualified researchers who meet the legal and ethical requirements governing data sharing. Access to the data will be provided by contacting the principal investigator of the study. This data sharing plan will be in effect for 5 years following the publication date
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: August 2025- August 2026
Access Criteria: Data requests should be sent via email to the principal investigator of the study. The email must include the planned research proposal and the institutional ethical approval document as attachments.
  Following a review of the request, a data sharing agreement will be signed with the researcher. This agreement will guarantee that the data will be used solely for the specified analyses and that confidentiality will be maintained.
  Upon the execution of the agreement, the de-identified data set and supporting documents (protocol, data collection forms, etc.) will be securely transferred to the researcher.

REFERENCES:
- [Background] Tucker WJ, Angadi SS, Gaesser GA. Excess Postexercise Oxygen Consumption After High-Intensity and Sprint Interval Exercise, and Continuous Steady-State Exercise. J Strength Cond Res. 2016 Nov;30(11):3090-3097. doi: 10.1519/JSC.0000000000001399. PMID 26950358